CLINICAL TRIAL: NCT06538298
Title: A Multimodal Exercise Program With Gamification (MEP+G) in Individuals With Parkinson Disease: a Pilot Randomized Controlled Trial
Brief Title: Title: A Multimodal Exercise Program With Gamification for Parkinson Disease (MEP+G)
Acronym: (MEP+G)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: California State University, Northridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY24-23
Record Dates: First submitted 2024-03-26; First posted 2024-08-05 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Multimodal Exercise; Gamification; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Exercise Program with Gamification (Experimental): The exercise program will be for 6 weeks, 3 days per week for 60 minutes per session and will consist of strengthening, balance, aerobic, flexibility, and use a computerized game to challenge thinking and reactions skills. The exercise program will also consist of non-contact boxing to improve strength, balance, and aerobic endurance.
  Each exercise session will be conducted by a licensed physical therapist. The format will consist of a 10-15-minute warm-up followed by 30 minutes of moderate to vigorous circuit training using boxing drills and a computerized game called SMARTfit. SMARTfit consists of a standing computer board that allows participants to touch, punch or kick it while playing a game. At the end of the 30 minutes, participants will complete a 10-15-minute cool-down consisting of core strengthening, posture training, and hip strengthening and stretching exercises. Participants will also be instructed to maintain their normal activities outside of the study intervention.
  Interventions: Other: Multimodal Exercise Program with Gamification
- Wait List Control (No Intervention): Participants randomly assigned to the wait list control group, will perform baseline testing and be instructed not to change their exercise habits. After 6 weeks participants will complete post-testing (described below) and be offered to be enrolled in the 6-week exercise group as described above. If participants decide to participate in the exercise group and still meet the inclusion and exclusion criteria, they will perform baseline testing, 6 weeks of exercise followed by another post-testing.

INTERVENTIONS:
Other: Multimodal Exercise Program with Gamification — A comprehensive exercise program for 3 days a week for 6 weeks that utilizes non-contact boxing and gamification at moderate to vigorous intensity.
  Arms: Multimodal Exercise Program with Gamification

SUMMARY:
In this pilot study the research will explore whether exercises and the outcome measures would be acceptable to conduct a more detailed research study. This 8 week pilot study will utilize a comprehensive exercise program that includes non-contact boxing along with computerized games for individuals with Parkinson Disease.

DETAILED DESCRIPTION:
Participates in the 6-week exercise group will be asked to perform the following three times per week for 6 weeks, with each session lasting 60 minutes: A multimodal group exercise program with approximately 3-5 other individuals with Parkinson's disease. The exercise program will consist of strengthening, balance, aerobic, flexibility, and the use of a computerized game to challenge participant's thinking and reactions skills. The exercise program will also consist of non-contact boxing (hitting punching bags) to improve strength, balance, and aerobic endurance. Each exercise session will be conducted by a licensed physical therapist who is trained in exercise programs using non-contact boxing (Certified Rock Steady Boxing Coach). Each exercise session will have the same format and exercises with only a slight variation. For example, all Monday classes will have a focus on strengthening, Wednesday classes will have a focus on balance and Friday classes will have a focus on power.

The format will consist of a 10-15-minute warm-up of stretching and exercises to gradually warm-up participant's muscles and increase heart rate. Following the warm-up, participates will complete 30 minutes of moderate to vigorous circuit training using boxing drills and a computerized game called SMARTfit. SMARTfit consists of a standing computer board that allows participants to touch, punch or kick it while playing a game i.e., hitting all the buttons that display a smiley face.

At the end of the 30 minutes, participants will complete a 10-15-minute cool-down consisting of core strengthening, posture training, and hip strengthening and stretching exercises. Participants will also be instructed to maintain their normal activities outside of the study intervention.

In the event participants missed any of the exercise sessions, a one-week "make up week" will be provided immediately following the 6-week intervention that participants can choose to attend.

Exercise Intensity will be monitored using a heart rate chest monitor (Myzone™). The Myzone™) heart rate monitor will allow the instructor/researcher to monitor heart rate during the exercise session via a computer screen and to evaluate exercise response after the session is completed to determine whether to increase or decrease the intensity. For the first two weeks, participants will be instructed to stay in the "moderate" range of intensity during the 30 minutes of circuit training. The following four weeks participants will be instructed to increase their effort to vigorous as assessed and determined by the instructor. Moderate intensity is defined as 70-80 percent of estimated maximum heart rate. Vigorous intensity is defined as 80-90 percent estimated maximum heart rate.

Estimated maximum heart rate is determined by: 208-.7 X age. Estimated maximum heart rate will be adjusted for participants on beta blockers or other blood pressure lowering medications (164-.7 X age).

At the end of each exercise session the instructor will complete the data sheet on the daily scripted exercise plan. For example, the instructor will document whether the participant was present, had any adverse events, able to complete the exercises as prescribed etc.

Wait List Control Group Participants randomly assigned to the wait list control group, will perform baseline testing and be instructed not to change their exercise habits. After 6 weeks participants will complete post-testing (described below) and be offered to be enrolled in the 6-week exercise group as described above. If participants decide to participate in the exercise group and still meet the inclusion and exclusion criteria, they will perform baseline testing, 6 weeks of exercise followed by another post-testing.

Week #10 (Post Testing): Participants will complete the same surveys and clinical measures as performed during for pre-testing. Post-testing will be approximately 60 minutes. Participants will also be provided qualitative and quantitative questions via an anonymous link and/or QR code to a Qualtrics survey pertaining to their experience and satisfaction with the program.

Quantitative questions will use a rating scale of 1-5 with 1= strongly agree; 2= somewhat agree; 3= neutral; 4; somewhat disagree; 5; strongly disagree. Questions will pertain to usefulness of the program, ease of use, burden of doing the exercises/testing, comprehensibility.

Qualitative questions will be open ended asking about most/least helpful components, met expectations, suggestions for improvement, perceived safety of doing the exercises and testing and intent to continue the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn and Yahr stages 1-3 disease as determined by primary care physician, neurologist, or movement disorder specialist
* diagnosis of idiopathic Parkinson's Disease
* ability to ambulate with or without an assistive device
* transportation to and from testing site
* ability to stand unassisted for 10 minutes
* stable on Parkinson's disease medications for 3 months as determined by physician
* medical clearance by their PCP, neurologist, or movement disorder specialist to participate in a moderate to vigorous exercise program.

Exclusion Criteria:

* other neurological disease other than Parkinson's disease
* having had deep brain stimulation within the past 3 months , as determined by their physician
* currently participating in a Rock Steady boxing program
* self-report participation in moderate to vigorous exercise greater than 60 minutes per week.

  * required

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-06-27 (Estimated)

PRIMARY OUTCOMES:
Fidelity of intervention | 21 months
  Participants completing exercises as prescribed: measured using the daily exercise plan as a "yes" or "no".
Intervention Adherence | 21 months
  Measured by daily exercise plan; instructors will indicate whether participant was present as a "yes" or "no"
Feasibility of Outcomes | 21 months
  Retention: number of participants who completed the entire program divided by total number who started; x 100 to determine the percentage of participants who completed the program.
Assessment of Data Collection | 21 months
  Data collection: measured using a pre-populated form and marked as a "yes" or "no" by the PI.
Assessment of Safety | 21 months
  Adverse events (i.e., falls): measured by the daily exercise plan as indicated by a numeric number and type of adverse event
Assessment of Participants Perception | 21 months
  Measured via Qualtrics survey asking participants "How satisfied were you in participating in this study" using an ordinal scale (0-4): (4)(strongly agree; (3)agree; (2)neutral; (1)disagree; (0)strongly disagree); with a higher score reflection increased satisfaction

SECONDARY OUTCOMES:
Balance | 21 months
  Measured via using the Mini Balance Evaluation System Test (Mini-BESTest): a series of subtests with a total score from 0-28 points; with a higher score indicating improved balance.
Gait | 21 months
  Measured via Functional Gait Assessment (FGA): series of subtests based out of score from 0- 30 points; with a higher score indicating improved postural stability while walking.
Physical Activity | 21 months
  Measured via International Physical Activity Questionnaire (IPAQ) based on minutes exercise per week with a higher number of minutes indicating increased physical activity
Gait Speed | 21 months
  Gait speed measured via 10 meters divided by number of seconds to determine gait speed of meters per second (m/s); a increased in m/s indicating improved gait speed.
Functional Strength | 21 months
  Functional strength measured by number of seconds required to perform 5 sit to stands (5TSTS) with a decrease in time indicating improved functional strength.
Cardiovascular Endurance | 21 Months
  Cardiovascular endurance measured by total number of feet walked within a 6 minute timeframe (6MWT); an increase number of steps indicating improved cardiovascular endurance.
Quality of life of Participants | 21 months
  Quality of life measured by Parkinson Disease Questionnaire: 39 (PDQ39) questions asking participants to rate various aspects of their condition using an ordinal scale: 0-4 (4)(Always, (3)Often, (2)Occasionally, (1)Sometimes, (0)Never; with a higher score indicating an increased quality of life
Disease Severity | 21 months
  Disease severity measured by the Movement Disorder Society Unified Parkinson DiseaseRating (MDS UPDRS); 18 items measured using an ordinal scale (0-4).0=none;1=slight;2=minimal;3; moderate;4=severe; with a lower score indicating less severity

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Bartlett, PhD, Principal Investigator — California State University, Northridge
Locations (1):
- Equilibrium Physical Therapy, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately upon completion and until publication
Access Criteria: Information will be shared upon request by the primary investigator.

REFERENCES:
- [Background] Schenkman M, Moore CG, Kohrt WM, Hall DA, Delitto A, Comella CL, Josbeno DA, Christiansen CL, Berman BD, Kluger BM, Melanson EL, Jain S, Robichaud JA, Poon C, Corcos DM. Effect of High-Intensity Treadmill Exercise on Motor Symptoms in Patients With De Novo Parkinson Disease: A Phase 2 Randomized Clinical Trial. JAMA Neurol. 2018 Feb 1;75(2):219-226. doi: 10.1001/jamaneurol.2017.3517. PMID 29228079
- [Background] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790
- [Background] El-Kotob R, Giangregorio LM. Pilot and feasibility studies in exercise, physical activity, or rehabilitation research. Pilot Feasibility Stud. 2018 Aug 14;4:137. doi: 10.1186/s40814-018-0326-0. eCollection 2018. PMID 30123527
- [Background] Landers MR, Ellis TD. A Mobile App Specifically Designed to Facilitate Exercise in Parkinson Disease: Single-Cohort Pilot Study on Feasibility, Safety, and Signal of Efficacy. JMIR Mhealth Uhealth. 2020 Oct 5;8(10):e18985. doi: 10.2196/18985. PMID 33016887
- [Background] Sangarapillai K, Norman BM, Almeida QJ. Boxing vs Sensory Exercise for Parkinson's Disease: A Double-Blinded Randomized Controlled Trial. Neurorehabil Neural Repair. 2021 Sep;35(9):769-777. doi: 10.1177/15459683211023197. Epub 2021 Jun 13. PMID 34121511
- [Background] Osborne JA, Botkin R, Colon-Semenza C, DeAngelis TR, Gallardo OG, Kosakowski H, Martello J, Pradhan S, Rafferty M, Readinger JL, Whitt AL, Ellis TD. Physical Therapist Management of Parkinson Disease: A Clinical Practice Guideline From the American Physical Therapy Association. Phys Ther. 2022 Apr 1;102(4):pzab302. doi: 10.1093/ptj/pzab302. PMID 34963139
- [Background] Langbroek-Amersfoort A, Schootemeijer S, Bouten L, Bloem BR, De Vries NM. Exercise Made Accessible: the Merits of Community-Based Programs for Persons with Parkinson's Disease. Curr Neurol Neurosci Rep. 2023 Nov;23(11):695-715. doi: 10.1007/s11910-023-01303-0. Epub 2023 Oct 4. PMID 37792207